CLINICAL TRIAL: NCT05861999
Title: A Phase IV Open-Label Study Evaluating the Effectiveness and Safety of Risdiplam Administered in Pediatric Patients With Spinal Muscular Atrophy Who Experienced a Plateau or Decline in Function After Gene Therapy
Brief Title: A Study Evaluating the Effectiveness and Safety of Risdiplam Administered in Pediatric Patients With Spinal Muscular Atrophy Who Experienced a Plateau or Decline in Function After Gene Therapy
Acronym: HINALEA 2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN44621; 2023-505161-81-00 (EU CTIS Number)
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Risdiplam (Experimental): Participants will receive risdiplam orally once daily for 72 weeks (Treatment Period). The Treatment Period will be followed by a 1-year Treatment Extension Period for a total study duration of 120 weeks (approximately 2.5 years) for each participant enrolled.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Risdiplam — Participants will receive risdiplam orally at the currently approved dose. The dose should be adapted for weight and age.
  Other Names: RO7034067

SUMMARY:
This is an open-label, single-arm, multicenter clinical study to evaluate the effectiveness and safety of risdiplam administered in pediatric participants with SMA and 2 SMN2 copies who previously received onasemnogene abeparvovec and experience a plateau or decline in function. Participants to be enrolled are children <2 years of age genetically diagnosed with SMA.

ELIGIBILITY:
Inclusion Criteria:

* <2 years of age at the time of informed consent
* Confirmed diagnosis of 5q-autosomal recessive SMA, including genetic confirmation of homozygous deletion or compound heterozygosity predictive of loss of function of the Survival of Motor Neuron 1 (SMN1) gene
* Confirmed presence of two SMN2 gene copies as documented through laboratory testing
* Administration of onasemnogene abeparvovec pre-symptomatically or post-symptomatically
* Has received onasemnogene abeparvovec for SMA no less than 13 weeks prior to enrollment
* If treated with risdiplam prior to onasemnogene abeparvovec, risdiplam treatment must not have exceeded 3 weeks and must be discontinued 1 day prior to onasemnogene abeparvovec administration.
* In the opinion of the investigator, has demonstrated a plateau or decline in function post-gene therapy (with a duration of 26 weeks or less) documented by 2 individual time points in the functions as follows: swallowing AND one additional function/ability (respiratory, motor function, other) per appropriate expectation.

Exclusion Criteria:

* Previous or current enrolment in investigational study prior to initiation of study treatment
* Any unresolved standard-of-care laboratory abnormalities per the onasemnogene abeparvovec prescribing information
* Concomitant or previous administration of an SMN2-targeting antisense oligonucleotide
* Concomitant or previous use of an anti-myostatin agent
* Participants requiring invasive ventilation or tracheostomy
* Presence of feeding tube and an OrSAT score of 0
* Hospitalization for pulmonary event within the last 2 months, or any planned hospitalization at the time of screening
* Any major illness requiring hospitalization within 1 month before the screening examination or any febrile illness within 1 week prior to screening and up to first dose administration.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Raw Score of Bayley Scales of Infant and Toddler Development - Third Edition (BSID-III) Gross Motor Score at 72 Weeks of Risdiplam Treatment | Baseline, Week 72
  The BSID-III is a standardized assessment commonly used to evaluate developmental functioning of infants and young children between 1 month and 42 months of age. The gross motor scale measures the movement of the limbs and torso. Items assess static positioning (e.g., sitting, standing); dynamic movement, including locomotion and coordination; balance; and motor planning. The gross motor scale consists of 72 items scored at 0 (unable to perform) or 1 (criteria for item achieved). A higher raw score indicates improvement.

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | Up to 120 weeks
Percentage of Participants With Serious Adverse Events | Up to 120 weeks
Percentage of Participants With Treatment Discontinuation Due to Adverse Events | Up to 120 weeks

OTHER OUTCOMES:
Change from Baseline in Bulbar/Swallowing Function Assessment as Measured by the Oral and Swallowing Abilities Tool (OrSAT) at 72 Weeks of Risdiplam Treatment and Over Time | From baseline up to Week 120
  The OrSAT is a validated assessment composed of a checklist of 12 questions assessing aspects of swallowing abilities thought to be clinically meaningful for a type 1 SMA population and developmentally appropriate for infants during the first months of life. Each item is graded with a score of 0 or 1, depending on the child's ability to perform the activity. As some items are age-dependent, the number of items to be used, and therefore the maximum score, changes with increasing age. In the infants younger than 6 months the maximum score is 7. For those between 6 and 9 months, maximum score is 10. For infants of 10 months or older, maximum total score is 12.
Change in Swallowing Function Assessment as Measured by the Pediatric Functional Oral Intake Scale (p-FOIS) Over Time | From baseline up to Week 120
  The p-FOIS is a 6-point scale that assesses feeding ability, 1= Nothing by mouth, 2= Tube dependent for all nutrition/hydration needs with minimal attempts at oral intake for experience and/or pleasure, 3= Tube dependent with consistent intake of food and/or fluid that meets some of the nutrition/hydration needs, 4= Total oral intake but special preparation required, e.g., thickened fluids, puréed diet (where not age-appropriate), 5= Total oral intake but requiring special conditions/modification, e.g., slow flow teat/side lying/pacing or specific food limitations, 6= Total, age-appropriate, oral intake with no restrictions. Higher score indicates higher level of function.
Change from Baseline in the Raw Score of BSID-III Gross Motor Score Over Time Under Risdiplam Treatment | From baseline up to Week 120
  The BSID-III is a standardized assessment commonly used to evaluate developmental functioning of infants and young children between 1 month and 42 months of age. The gross motor scale measures the movement of the limbs and torso. Items assess static positioning (e.g., sitting, standing); dynamic movement, including locomotion and coordination; balance; and motor planning. The gross motor scale consists of 72 items scored at 0 (unable to perform) or 1 (criteria for item achieved). A higher raw score indicates improvement.
Percentage of Participants With a Gross Motor Index Between 80-109 as Measured by the Peabody Developmental Motor Scale, Third Edition (PDMS-3) at 72 Weeks of Risdiplam Treatment and Over Time | From baseline up to Week 120
  The PDMS-3 is used to assess gross- and fine-motor skills in children from birth to 5 years. The PDMS-3 has 3 composite scores: Total Motor (combined scores of the core subtests) and two domain composites (Gross Motor and Fine Motor). By combining the results of subtests, these composite scores are considered to have stronger and better indexes of performance and, therefore, more reliable and valid than the subtests. Score for composite indexes range from <70 (impaired or delayed) to >129 (gifted or very advanced). Score of 80-89 indicate below average and 90-109 indicate average skills.
Percentage of Participants With a Fine Motor Index Between 80-109 as Measured by the PDMS-3 at 72 Weeks of Risdiplam Treatment and Over Time | From baseline up to Week 120
  The PDMS-3 is used to assess gross- and fine-motor skills in children from birth to 5 years. The PDMS-3 has 3 composite scores: Total Motor (combined scores of the core subtests) and two domain composites (Gross Motor and Fine Motor). By combining the results of subtests, these composite scores are considered to have stronger and better indexes of performance and, therefore, more reliable and valid than the subtests. Score for composite indexes range from <70 (impaired or delayed) to >129 (gifted or very advanced). Score of 80-89 indicate below average and 90-109 indicate average skills.
Change in World Health Organization (WHO) Motor Milestone Achievement at 72 Weeks of Risdiplam Treatment and Over Time | From baseline up to Week 120
  The WHO motor milestones evaluate gross motor development and comprise the time windows of achievement for six gross motor milestones based on data derived from the WHO Multicenter Growth Reference Study (MGRS). The six gross motor milestones are as follows: sitting without support, hands-and-knees crawling, standing with assistance, walking with assistance, standing alone, and walking alone. A yes response indicates that the participant reached a particular development milestone.
Percentage of Participants With Improvement or No Change in Respiratory Illness as Assessed by Clinical Global Impression of Change (CGI-C) | As per respiratory event on Day 10 and Day 20 postevent (up to Week 120)
  In a case of respiratory illness during the study, a range of clinical domain level items will be completed by the investigator, as needed. The CGI-C is a single item measure of change using seven response options: "Very much improved," "Much improved," "Minimally improved," "No change," "Minimally worse," "Much worse," and "Very much worse."
Percentage of Participants Within 3rd Percentile of Normal Range for Weight-to-Age at 72 Weeks of Risdiplam Treatment and Over Time | From baseline up to Week 120
Percentage of Participants Within 3rd Percentile of Normal Range for Length/Height-to-Age at 72 Weeks of Risdiplam Treatment and Over Time | From baseline up to Week 120
Percentage of Participants Within 3rd Percentile of Normal Range for Weight-to-Length/Height at 72 Weeks of Risdiplam Treatment and Over Time | From baseline up to Week 120
Number of Respiratory-Related Hospitalizations During the 72-Week Risdiplam Treatment and Over Time | Up to 120 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (10):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Valley Children's Hospital, Madera, California
  - Stanford Univ Medical Center, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - University of Florida Pediatrics, Gainesville, Florida
  - Children's Healthcare of Atlanta Center for Advanced Pediatrics, Atlanta, Georgia
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children'S Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Children's Hospital of the King's Daughter, Norfolk, Virginia
- Germany (2):
  - Charité - Universitätsmedizin Berlin SPZ Abteilung Neuropaediatrie, Berlin
  - UKGM Standort Gießen, Giessen
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - Sourasky MC, Dana-Dwek Children's Hospital, Tel Aviv
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
- Sidra Medicine, Al Rayyan, Qatar
- Great Ormond Street Hospital For Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This clinical trial evaluates treatment of a rare genetic disease in a small cohort of participants. No data is planned to be shared in order to protect and maintain participant privacy/confidentiality.